CLINICAL TRIAL: NCT05634382
Title: Endovascular Thrombectomy With and Without Intravenous Thrombolysis for Large Vessel Anterior Circulation Stroke in Extended Time Window
Brief Title: Endovascular Thrombectomy With and Without Intravenous Thrombolysis in Extended Time Window
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HOPE-BRIDGING
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous thrombolysis bridging with endovascular thrombectomy (Experimental)
  Interventions: Drug: Intravenous thrombolysis agents; Procedure: endovascular thrombectomy
- Direct endovascular thrombectomy without intravenous thrombolysis (Active Comparator)
  Interventions: Procedure: endovascular thrombectomy

INTERVENTIONS:
Drug: Intravenous thrombolysis agents — Intravenous thrombolysis with recombinant tissue-type plasminogen activator (rt-PA，alteplase) or TNK-tPA (Tenecteplase，Metalyse)
  Arms: Intravenous thrombolysis bridging with endovascular thrombectomy
Procedure: endovascular thrombectomy — endovascular mechanical thrombectomy with nonspecific device

SUMMARY:
The primary hypothesis being tested in this trial is that ischemic stroke patients in large vessel occlusion of anterior circulation at 4.5 - 9 hours post onset of stroke will have improved clinical outcomes when given endovascular thrombectomy with intravenous thrombolysis compared with that of given direct endovascular thrombectomy alone.

DETAILED DESCRIPTION:
A number of multicenter randomized controlled trials have provided evidence supporting the application of endovascular therapy for acute ischemic stroke with anterior circulation large vessel occlusion. However, whether intravenous thrombolysis is necessary before endovascular therapy is still controversial. The combined trial data (including DEVT, DIRECT-MT, MR-CLEAN NO-IV and SKIP) assessing direct mechanical thrombectomy versus bridging therapy showed no difference in improving good functional outcome. However, a recent observational cohort study of 15832 patients treated with EVT, intravenous alteplase treatment was associated with better in-hospital survival and functional outcomes after adjusting for other covariates.

The 2019 AHA/ASA guidelines for the early management of patients with ischemic stroke states that mechanical thrombectomy is recommended for patients with anterior circulation large vessel occlusion within 6-24 hours of last known normal who meet the DWAN or DEFUSE-3 criteria (level I recommendation, level A evidence). The DEFUSE 3 perfusion-infarction core mismatch criteria is: core infarct volume <70mL, ischemic penumbra volume >15mL, and hypoperfusion volume/core infarct volume >1.8. Intravenous thrombolytic therapy is recommended for patients with ischemic stroke within 4.5 hours of onset. A meta-analysis of three randomized controlled trials recently published in the Lancet found that ischemic stroke at 4.5 to 9 hours of onset or wake stroke was consistent with a core infarct volume <70mL, a penumbra volume >10mL, and a hypoperfusion volume/core infarct volume >1.2. Benefit from intravenous thrombolytic therapy (3 month mRS 0-1 ratio, thrombolytic vs non-thrombolytic: 36% vs 29%). It was also strongly recommended by 2021 ESO guidelines on intravenous thrombolysis for acute ischemic stroke.

For these reasons the investigators hypothesize that endovacular thrombectomy bridging with intravenous thrombolysis is superior to direct thrombectomy in patients of stroke at 4.5 to 9 hours, guided with perfusion imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patient/Legally Authorized Representative has signed the Informed Consent form
2. Age ≥ 18
3. Clinical signs consistent with an acute ischemic stroke
4. Neurological deficit with a NIHSS of ≥ 6 (deficits judged to be clearly disabling at presentation)
5. Patient is eligible for intravenous thrombolysis
6. Patient is eligible for endovascular treatment
7. Randomization no later than 8 hours 45 minutes after stroke symptom onset and initiation of IV t-PA must be started within 9 hours of stroke symptoms onset (for stroke with unknown time of onset, the midpoint of the time last known to be well and symptom recognition time)
8. ICA or MCA-M1 occlusion (carotid occlusions can be cervical or intracranial; with or without tandem MCA lesions) by MRA or CTA (including the reconstructed CTA derived from CTP). And target Mismatch Profile on CT perfusion or MRI (ischemic core volume is < 70 ml, mismatch ratio is >/= 1.8 and mismatch volume is >/= 15 ml)
9. Core-infarct volume of Alberta Stroke Program Early CT Score (ASPECTS) ≥ 6 based on baseline CT or MR imaging (MRI) (a region has to have diffusion abnormality in 20% or more of its volume to be considered MR-ASPECTS positive)

Exclusion Criteria:

1. Acute intracranial hemorrhage
2. Any contraindication for IV t-PA
3. Pre-treatment with IV t-PA
4. Pregnancy or lactating women. A negative pregnancy test before randomization is required for all women with child-bearing potential.
5. Known (serious) sensitivity to radiographic contrast agents, nickel, titanium metals, or their alloys
6. Known current participation in a clinical trial (investigational drug or medical device)
7. Renal insufficiency as defined by a serum creatinine > 2.0 mg/dl (or 176.8 µmol/l) or glomerular filtration rate (GFR) < 30 mL/min or requirement for hemodialysis or peritoneal dialysis
8. Severe comorbid condition with life expectancy less than 90 days at baseline
9. Known advanced dementia or significant pre-stroke disability (mRS score of ≥2)
10. Foreseeable difficulties in follow-up due to geographic reasons (e.g. patients living abroad)
11. Comorbid disease or condition that would confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments
12. Subject currently uses or has a recent history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than four alcoholic drinks per day).
13. Known history of arterial tortuosity, pre-existing stent, other arterial disease and/or known disease at the femoral access site that would prevent the device from reaching the target vessel and/or preclude safe recovery after MT
14. Radiological confirmed evidence of mass effect or intracranial tumor (except small meningioma)
15. Radiological confirmed evidence of cerebral vasculitis
16. CTA or MRA evidence of carotid artery dissection
17. Evidence of additional distal intracranial vessel occlusion in another territory (i.e. A2 segment of anterior cerebral artery or M3, M4 segment of MCA) on initial NCCT/MRI or CTA/MRA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2022-12-03 (Actual); Primary Completion 2024-11-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Good clinical outcome | 90 days after randomization
  Score in modified Rankin Scale (mRS) ≤ 2 (mRS is short for modified ranking score, with minimum value of 0 and maximum value of 6. Higher score means a worse outcome.)

SECONDARY OUTCOMES:
Mortality | 90 days after randomization
  Mortality due to any cause
Modified Rankin Scale (mRS) shift analysis | day 0 and 90 days after randomization
  (mRS is short for National Institute of health stroke scale, with minimum value of 0 and maximum value of 6. Higher score means a worse outcome.)
National Institute of Health Score Scale (NIHSS) | day 0 and day 1 after randomization
  (NIHSS is short for modified ranking score, with minimum value of 0 and maximum value of 42. Higher score means a worse outcome.)
Thrombolysis in Cerebral Infarction (TICI) scale | day 0 and day 1 after randomization
  TICI is for "Thrombolysis in cerebral Infarction", with minimum value of 0 and maximum value of 3. Higher score means a better reperfusion state.
Serious adverse events | day 0 until 90 days after randomization
  Leading to death or prolonged hospitalisation
Intracranial hemorrhage | day 1 after randomization
  Hemorrhagic finding on CT or MRI
Quality of life assessed by questionnaire | 90 days after randomization
  Include but not limited to the Barthelindex of ADL, which is the abbreviation of " activities of daily living", with minimum value of 0 and maximum value of 100. Higher score means a worse outcome.
Overall costs incurred during hospitalisation | 90 days after randomization
  include charges and expenses of every description

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, Professor, Principal Investigator — Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China